CLINICAL TRIAL: NCT07274722
Title: Influence of Control Deprivation on the Use of the Analytical Cognitive Style in Anorexic Subjects
Acronym: PriCo-SCASA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Collaborators: Centre de Recherches sur la Cognition et l'Apprentissage (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-A00826-39
Record Dates: First submitted 2025-06-03; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Control Deprivation (Experimental)
  Interventions: Other: Cognitive Control Deprivation Task

INTERVENTIONS:
Other: Cognitive Control Deprivation Task — The investigators will measure the reaction time to the detection of a stimulus requiring analytical information processing compared with the time required to detect a stimulus requiring global information processing. These measurements will be carried out before and after a cognitive control deprivation experiment, which will be used to activate a need for control in the experimental context. The two measures will then be compared to examine the changes that occur after the deprivation of control.

SUMMARY:
The use of an analytical cognitive style is a specific feature of anorexia nervosa and is thought to contribute to the maintenance of the disorder, in particular by encouraging fragmented body perception and a focus on certain parts of the body to the detriment of overall harmony and coherence. The need for control has also been described as an important element in the pathology. At the same time, some authors have shown that, outside of any pathology, recourse to the analytical cognitive style could respond to a need to restore control and, in turn, improve the feeling of control. However, at present, no causal relationship has been demonstrated between the feeling of loss of control and the analytical cognitive style in anorexia nervosa. However, such a relationship would enable us to gain a better understanding of the underlying mechanisms of the disorder and to better target the treatment of patients.

ELIGIBILITY:
Inclusion Criteria:

* Be undergoing treatment at Centre Hospitalier Laborit (CHL) or Centre Hospitalier Universitaire (CHU) de Poitiers for an Eating Disorder (ED) of the Anorexia Nervosa type.
* Patients must meet the diagnostic criteria for Anorexia Nervosa according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5; American Psychiatric Association, APA, 2013), or present a sub-clinical symptomatology requiring treatment:

(A) Restriction of energy intake relative to requirements, leading to a significantly low body weight, taking into account age, sex, developmental stage, and physical health; (B) Intense fear of gaining weight or becoming fat, or persistent behavior that interferes with weight gain, even when at a significantly low weight; (C) Disturbance in the way body weight or shape is experienced, undue influence of body weight or shape on self-esteem, or persistent lack of recognition of the seriousness of the current low body weight.

Exclusion Criteria:

* Objection of the referring therapist
* Currently receiving cognitive remediation targeting mental flexibility and central coherence
* Body Mass Index (BMI) less than 14
* Inability to understand instructions in French
* Visual impairment or dyslexia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Reaction time | Baseline (before cognitive control deprivation) and immediately post-task (after cognitive control deprivation on Day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France